CLINICAL TRIAL: NCT05545865
Title: Preclinical Trials to Determine the Range of Chardonnay Mark Intake for Improved Metabolic and Vascular Response.
Brief Title: Chardonnay Marc and Vascular Response
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 1810396
Record Dates: First submitted 2022-09-09; First posted 2022-09-19 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Cardiovascular Diseases; Vascular Dilation; Oxidative Stress
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Acute crossover design
Who Masked: Participant, Investigator
Masking Description: Low and High flavanol cocoa will be provided in coded packaging.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Low Flavanol Cocoa Powder (Placebo Comparator): 12 g of Low Flavanol Cocoa Powder (30 mg of cocoa flavanols) provided as a beverage mixed in water
  Interventions: Other: High Flavanol Cocoa Powder; Other: Vine to Bar Chocolate - 2 servings; Other: Vine to Bar Chocolate - 1 serving
- High Flavanol Cocoa Powder (Experimental): High Flavanol Cocoa Powder (435 mg of flavanols) will be provided as a beverage mixed in water.
  Interventions: Other: Low Flavanol Cocoa Powder; Other: Vine to Bar Chocolate - 2 servings; Other: Vine to Bar Chocolate - 1 serving; Other: Vine to Bar Chocolate covered almonds
- Two Servings of Vine to Bar Chocolate (Experimental): Two servings (60g, 6 pieces) of Vine to Bar Chocolate providing both cocoa flavanols and Chardonnay marc.
  Interventions: Other: Vine to Bar Chocolate - 1 serving; Other: Vine to Bar Chocolate covered almonds
- One Serving of Vine to Bar Chocolate (Experimental): A single serving (30g, 3 pieces) of Vine to Bar Chocolate providing both cocoa flavanols and Chardonnay marc.
  Interventions: Other: Low Flavanol Cocoa Powder; Other: High Flavanol Cocoa Powder; Other: Vine to Bar Chocolate - 2 servings; Other: Vine to Bar Chocolate covered almonds
- Vine to Bar Chocolate covered Almonds (Experimental): 11 pieces (45g) of Vine to Bar Chocolate providing both cocoa flavanols and Chardonnay marc, with almonds
  Interventions: Other: Vine to Bar Chocolate - 2 servings; Other: Vine to Bar Chocolate - 1 serving

INTERVENTIONS:
Other: Low Flavanol Cocoa Powder — Measure the response 2 and 6 hours post low flavanol cocoa intake
  Arms: High Flavanol Cocoa Powder; One Serving of Vine to Bar Chocolate
Other: High Flavanol Cocoa Powder — Measure the response 2 and 6 hours post high flavanol cocoa intake
  Arms: Low Flavanol Cocoa Powder; One Serving of Vine to Bar Chocolate
Other: Vine to Bar Chocolate - 2 servings — Measure the response 2 and 6 hours post chocolate intake
  Arms: High Flavanol Cocoa Powder; Low Flavanol Cocoa Powder; One Serving of Vine to Bar Chocolate; Vine to Bar Chocolate covered Almonds
Other: Vine to Bar Chocolate - 1 serving — Measure the response 2 and 6 hours post chocolate intake
  Arms: High Flavanol Cocoa Powder; Low Flavanol Cocoa Powder; Two Servings of Vine to Bar Chocolate; Vine to Bar Chocolate covered Almonds
Other: Vine to Bar Chocolate covered almonds — Measure the response 2 and 6 hours post chocolate covered almond intake
  Arms: High Flavanol Cocoa Powder; One Serving of Vine to Bar Chocolate; Two Servings of Vine to Bar Chocolate

SUMMARY:
This study aims to obtain data on the potential influence of Vine to Bar product(s) containing Chardonnay marc on cardiometabolic health. These initial studies will inform the design and timing of data collection for future dietary intervention trials that will examine the influence of Chardonnay marc intake on outcomes/biomarkers of both cardiometabolic health and the gut microbiome. This includes collecting data on the potential differences in response to the products based on the unique food matrix for each of the products that will be tested. Moreover, as there is a paucity of data on the influence of cocoa flavanol intake on vascular function beyond 4 hours post intake, the response of the selected outcomes will be assessed after 6 hours of flavanol intake. This is a time point that captures the increased circulating presence of microbial derived flavanol metabolites.

DETAILED DESCRIPTION:
The current set of trials will be of an acute (single intake, followed over 6 hours) that examines the postprandial response of individuals to the products. These preclinical trials will be conducted in the same individuals in an crossover design in order to limit individual variability, and keep the numbers small (5 individuals maximum), but still be able to assess the response to the different products.

ELIGIBILITY:
Inclusion Criteria:

* Screening or Visit 1 Reactive Hyperemia Index (RHI; EndoPAT 2000) < 2.0
* Subject is willing and able to comply with the study protocols.
* Subject is willing to participate in all study procedures
* BMI 25.0 - 35 kg/m2

Exclusion Criteria:

* BMI ≥ 35 kg/m2
* Indivduals that weight less than a 110 lbs
* Donation of blood within the previous 30 days
* Visit 1 Reactive Hyperemia Index (RHI; EndoPAT 2000) ≥ 2.0
* 1 ug/ml and 3 ug/ml collagen screening maximal platelet aggregatory response of < 65%.
* Platelet counts < 150,000 / ul
* Anemia, which includes self report, or a screening hemoglobin and hematocrit that is less than the normal reference range or as diagnosed by study physician upon review of complete blood cell count reports.
* Dislike or allergy for nuts, cocoa or grape products
* Self-reported use of daily anticoagulation agents including aspirin, NSAIDs
* Vegan, Vegetarians, food faddists or those consuming a non-traditional diet
* Fruit consumption ≥ 3 cups/day
* Vegetable consumption ≥ 4 cups/day
* Nut intake ≥ 2 servings/ week
* Coffee/tea ≥ 3 cups/day
* Dark chocolate ≥ 3 oz/day
* Self-reported restriction of physical activity due to a chronic health condition
* Self-reported chronic/routine high intensity exercise
* Self-reported diabetes
* Blood pressure ≥ 140/90 mm Hg
* Self-reported renal or liver disease
* Self-reported heart disease, which includes cardiovascular events and stroke
* Peripheral artery disease, Raynaud's syndrome
* Inability to properly place or wear the PAT probes or abnormal measurements on pre- screening PAT
* Self-reported cancer within past 5 years
* Self-reported malabsorption
* Currently taking prescription drugs or supplements.
* Supplement use or unwillingness to stop any supplement use, including herbal, plant or botanical, fish oil, oil supplements a month prior to study enrollment.
* Indications of substance or alcohol abuse within the last 3 years
* smoking, vaping, cannabis use
* Current enrollee in a clinical research study.

Ages: 30 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-08-24 (Estimated); Study Completion 2025-08-24 (Estimated)

PRIMARY OUTCOMES:
Framingham Reactive Hyperemia Index (fRHI) | 6 hours
  measurement of microvascular function using peripheral arterial tonometry (EndoPAT2000)

SECONDARY OUTCOMES:
Platelet aggregation | 6 hours
  Platelet aggregation after collagen activation will be assessed using platelet aggregometry
soluble NADPH oxidase | 6 hours
  measure of oxidative stress
Glucose | 6 hours
  Plasma glucose will be measured
Insulin | 6 hours
  Serum insulin levels will be measured
Total nitrate | 6 hours
  circulating levels of nitrate

CONTACTS AND LOCATIONS:
Overall Officials: Carl L Keen, Principal Investigator — Distinguished Professor Emeritus of Nutrition
Locations (1):
- Academic Surge, University of California, Davis, Davis, California, United States

IPD SHARING:
Plan to Share IPD: No